CLINICAL TRIAL: NCT02859883
Title: Evaluation of Oesogastroduodenoscopy With Vision to 245 ° (Full Spectrum Endoscopy) to View the Main Disc and Accessory
Acronym: FUSE-TM-Duo
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: FUSE-TM-Duodénum-IPC 2015-001
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-04

CONDITIONS: Adenoma of the Accessory Papilla; Ampulloma of the Accessory Papilla

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: gastroscope FUSE™ — All patients undergoing a diagnostic gastroscopy are eligible. Using the FUSE endoscope with side screen, the duodenal and accessory papilla are monitored. Data are collected by each operator. Clinical examination of patients is performed before they leave the centre.

SUMMARY:
The monitoring and prognosis of patients with familial polyposis adenomatous rests on analysis of the transitional mucosa at the anal margin and especially on the tracking, characterization and resection of lesions of dysplasia type of high grade at the duodenal level, after total proctocolectomy. Currently, endoscopes with axial or lateral vision are used. The FUSE technology allows the simplification or even the improvement of patient surveillance with a 245° vision (versus150° in case of classical gastroscope). The use of a second screen to enlarge the field of view may allow both analysis of duodenum and the main and accessory papilla with one single endoscope and to decrease the number of omitted lesions .

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible to any upper gastrointestinal endoscopy diagnostic

Exclusion Criteria:

* History of duodenal or gastric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient eligible to any upper gastrointestinal endoscopy diagnostic
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 day
  Visualization of minor and major papilla Absence of necessity to change endoscope for viewing and / or for biopsies

SECONDARY OUTCOMES:
Number of patient with treatment-related serious adverse events | 5 day
  Evaluated serious advers events are mainly perforation, severe bleeding, acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe RATONE, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches du Rhone, France

REFERENCES:
- [Background] Gralnek IM, Segol O, Suissa A, Siersema PD, Carr-Locke DL, Halpern Z, Santo E, Domanov S. A prospective cohort study evaluating a novel colonoscopy platform featuring full-spectrum endoscopy. Endoscopy. 2013 Sep;45(9):697-702. doi: 10.1055/s-0033-1344395. Epub 2013 Aug 12. PMID 23939509
- [Background] Gralnek IM, Siersema PD, Halpern Z, Segol O, Melhem A, Suissa A, Santo E, Sloyer A, Fenster J, Moons LM, Dik VK, D'Agostino RB Jr, Rex DK. Standard forward-viewing colonoscopy versus full-spectrum endoscopy: an international, multicentre, randomised, tandem colonoscopy trial. Lancet Oncol. 2014 Mar;15(3):353-60. doi: 10.1016/S1470-2045(14)70020-8. Epub 2014 Feb 20. PMID 24560453
- [Background] Moussata D, Napoleon B, Lepilliez V, Klich A, Ecochard R, Lapalus MG, Nancey S, Cenni JC, Ponchon T, Chayvialle JA, Saurin JC. Endoscopic treatment of severe duodenal polyposis as an alternative to surgery for patients with familial adenomatous polyposis. Gastrointest Endosc. 2014 Nov;80(5):817-25. doi: 10.1016/j.gie.2014.03.012. Epub 2014 May 6. PMID 24814771